CLINICAL TRIAL: NCT05170867
Title: The Impact of Hafnia Alvei on Weight Loss and Glycaemic Control After Bariatric Surgery - A Randomized, Triple-blind, Controlled Trial
Brief Title: The Impact of Hafnia Alvei on Weight Loss and Glycaemic Control After Bariatric Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Academia CUF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RESTART
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Gut microbiota; Probiotics
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Two capsules of Hafnia alvei HA4597™ probiotic/day (5 x 107 CFU/day) for 90 days
  Interventions: Dietary Supplement: Hafnia alvei HA4597™
- Placebo group (Placebo Comparator): Two identical capsules of placebo/day for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Hafnia alvei HA4597™ — One capsule of probiotic supplement, twice a day, to be taken with water, during each breakfast and lunch (approx. 5 minutes after starting eating), for 90 days. Two capsules of the dietary supplement contain 5x107 CFU of Hafnia alvei HA4597™, 5 mg of zinc and 20 μg of chromium.
  Arms: Probiotic group
Other: Placebo — One capsule of placebo, twice a day, to be taken with water, during each breakfast and lunch (approx. 5 minutes after starting eating), for 90 days. Two capsules of the placebo contain 5 mg of zinc and 20 μg of chromium.
  Arms: Placebo group

SUMMARY:
This study aims to investigate the effects of Hafnia alvei HA4597 TM supplementation on weight loss and glycemic control after bariatric surgery. Patients undergoing Roux-en-Y gastric bypass will receive probiotics or placebo, twice a day, for 90 days, one month after surgery. Outcomes will be measured at baseline, and 3, 6, 9 and 12 months after the surgery.

DETAILED DESCRIPTION:
Gut microbiota dysbiosis is associated with the pathophysiology of obesity. Bariatric surgery is an effective treatment for obesity that induces changes in the gut microbiota. However, recent studies indicate that the gut microbiota is not fully restored after bariatric surgery which may limit the potential of the surgery to achieve metabolic control and maintain weight loss. Thus, modulating the gut microbiota with probiotics after bariatric surgery could be an effective strategy to improve the success of the surgery.

This study aims to investigate the effects of Hafnia alvei HA4597 TM supplementation on weight loss and glycemic control after bariatric surgery. Patients undergoing Roux-en-Y gastric bypass will receive probiotics or placebo, twice a day, for 90 days, one month after surgery. Outcomes will be measured at baseline, and 3, 6, 9 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years
* BMI ≥35 kg/m2 and at least one severe obesity-related complications, or BMI ≥40 kg/m2
* Undergoing Roux-en-Y gastric bypass
* Willing to take a probiotic/placebo supplement twice a day for 60 days
* Willing and able to provide written informed

Exclusion Criteria:

* Intake of antibiotics and/or probiotics in the previous 12 weeks
* Weight change >5% in the previous 12 weeks
* Diagnosis of gastrointestinal disease or other significant illness
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in percentage of excess weight loss from baseline.
HbA1c | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in HbA1c levels (%) from baseline.

SECONDARY OUTCOMES:
Gut microbiota | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in gut microbiota from baseline. Bacterial DNA will be extracted from faecal samples. 16S rRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Gastrointestinal quality of life | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in gastrointestinal quality of life by the Gastrointestinal Quality of Life Index (GIQLI) questionnaire from baseline. The GIQLI is a 36 -item questionnaire and consists of 5 different subscales. The total score is calculated as the sum of the 36 items each ranged from 0 to 4. The final score range from 0 to 144 points (lower scores indicate more unfavorable conditions).
Caseinolytic protease B | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in caseinolytic protease B (pM) from baseline.
Gut microbiota metabolites | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in short-chain fatty acids (acetate, propionate and butyrate) concentrations (mg/mL) from baseline. Short-chain fatty acids will be measured by targeted metabolomics.
Fasting blood glucose | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in fasting blood glucose levels (mg/dL) levels from baseline.
Insulin | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in insulin levels (μU/mL) levels from baseline.
C-peptide | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in c-peptide levels (ng/mL) levels from baseline.
Total cholesterol | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in total cholesterol levels (mg/dL) from baseline.
HDL cholesterol | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in high-density lipoprotein (HDL) cholesterol (mg/dL) levels from baseline.
LDL cholesterol | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in low-density lipoprotein (LDL) cholesterol (mg/dL) levels from baseline.
Triacylglycerides | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in triacylglycerides (mg/dL) levels from baseline.
Body fat mass | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in percentage of body fat mass from baseline.
Free fat mass | At visit 1 (Baseline), visit 2 (3 months after bariatric surgery), visit 3 (6 months after bariatric surgery), visit 4 (9 months after bariatric surgery), visit 5 (12 months after bariatric surgery).
  Changes in free fat mass (kg) from baseline.
Proportion of subjects losing more than 50% of baseline excess weight | At visit 1 (Baseline), visit 5 (12 months after bariatric surgery).
  Percentage of subjects losing >50% of baseline excess weight from baseline to visit 5 (12 months after bariatric surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School|Faculdade de Ciências Médicas, Universidade NOVA de Lisboa, Lisbon, Portugal

REFERENCES:
- [Derived] Ismael S, Vaz C, Durao C, Silvestre MP, Calhau C, Teixeira D, Marques C. The impact of Hafnia alvei HA4597 on weight loss and glycaemic control after bariatric surgery - study protocol for a triple-blinded, blocked randomized, 12-month, parallel-group, placebo-controlled clinical trial. Trials. 2023 May 29;24(1):362. doi: 10.1186/s13063-023-07383-0. PMID 37248499